CLINICAL TRIAL: NCT06734624
Title: Using Blood and Stool Samples From Patients With Blood Cancer and/or Haemophagocytic Lymphohistiocytosis to Study the Influence of Host Microbial Factors on Toxicity and Survival
Brief Title: The Microbiome in Blood Cancer and HLH
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 24059
Record Dates: First submitted 2024-11-11; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Haemophagocytic Lymphohistiocytosis
Keywords: Microbiome; DLBCL; FL; HLH
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and stool samples at three timepoints for each patient enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diffuse Large B-cell lymphoma (DLBCL): Patents with DLBCL receiving CART or Bispecific antibody treatment
- Follicular lymphoma (FL): Patents with newly diagnosed FL, or FL receiving CART or Bispecific antibody treatment
- Haemophagocytic lymphohistiocytosis (HLH): Patients who develop HLH with any underlying trigger factor.

SUMMARY:
The bacteria and viruses in the bowel (gut microbiota; GM) have powerful effects on the immune system. GM changes are seen in patients with auto-immune diseases, where the immune system attacks normal tissues, and cancer, and for those with some forms of blood cancer, and appears to affect both responses to, and side-effects of treatment. The investigators want to examine the GM and the associated small molecules (metabolites) in adults with different forms of blood cancer, particularly those undergoing immunotherapy, those with have newly diagnosed follicular lymphoma, and also those with a severe hyperinflammatory disorder which causes problems similar to sepsis called Haemophagocytic lymphohistiocytosis (HLH), which is also often caused by an underlying lymphoma. The investigators want to collect blood and stool samples from patients and use the results of tests already performed in the NHS as well as recording how well patients responded to treatment. The samples will be used to identify novel targets within the GM and associated metabolites which contribute to side effects of, or response to immunotherapy, or are responsible for causing HLH which can be targeted to make treatment better tolerated. For patients with newly diagnosed indolent lymphoma the aim is to see if there are differences which may account for patients needing early or late treatment, or no treatment ever.

DETAILED DESCRIPTION:
Introduction Immuno-therapy in the form of bispecific antibodies (BiSp) and chimeric antigen receptor T-cell (CAR-T) therapy have resulted in a paradigm shift in treatment for both aggressive and indolent B-cell lymhomas such as diffuse large B-cell lymphom and (DLBCL) and follicular lymphoma (FL). Immunotherapy utilises the patient's own immune system to help fight their diseases. Despite transformative results, CAR-T continues to have limitations in terms of both efficacy and adverse events, with a toxicity profile characterised by T-cell proliferation and over-activation primarily in the form of cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) with frequent intensive care admissions. CRS is a non-antigen-specific toxicity that occurs as a result of high-level immune activation, while the underlying mechanism driving ICANS is not fully understood, but is thought to relate to the release of inflammatory cytokines increasing vascular permeability, endothelial activation and leading blood-brain barrier breakdown. Similar toxicities are seen with BiSp although mitigation in the form of step up dosing and corticosteroid prophylaxis means these are somewhat less than that seen with CAR-T.

Haemophagocytic Lymphohistiocytosis (HLH) is a rare and often lethal hyper-inflammatory syndrome induced by aberrantly activated macrophages and cytotoxic T-cells. Patients develop fever, cytopenias and haemophagocytosis which may rapidly develop into multi-organ failure, akin to CRS. In general, infants tend to have inherited T- and NK-cell defects impairing cytotoxic function, younger adults have underlying acute viral infections and autoimmunity while older adults are those most likely to suffer from underlying cancer and have extremely poor outcomes

Over the past decade, a body of literature has emphasised interplay between the gut microbiota (GM), the immune system and the gut-brain axis. Compositional and functional changes in the GM (gut dysbiosis) may result in expansion of pro-inflammatory pathobionts with potential to enter the blood circulation, triggering cytokine signalling, as well as loss of normally residing microbiota or general loss of diversity. Host-gut microbiota interactions are mediated by small molecule metabolites, and dysbiosis may lead to alterations in innate and adaptive immunity, including regulatory T-cell generation and NK-cell function. Recent studies suggest dysbiosis to be associated with inferior outcomes and greater toxicity following CAR-T cell therapy. A retrospective study examining reported broad spectrum antibiotic therapy prior to CAR-T to be associated with worse survival and increased neurotoxicity, with the presence of Clostridia species associated with complete response. A further study found significant correlations between baseline Bifi dobacterium longum abundance and survival, and developed an algorithm predicting responders based on Bacteroides, Ruminococcus, Eubacterium, and Akkermansia abundance. These studies suggest the GM is intertwined with outcomes following CAR T-cell therapy but the mechanism and pathophysiology are not yet known. To date, there is no data regarding the GM and BiSp responses or immune related toxicities, or outcomes following a diagnosis of HLH.

In order to understand the effects of both the GM and the host immune system on blood cancer in general as well as outcomes and toxicities of immunotherapies in blood cancer and HLH, the investigators plan to prospectively collect stool and blood samples from patients undergoing treatment at multiple time-points. These samples will be used to characterise changes in GM and faecal metabolites, aiming to identify novel inflammatory pathogenic pathways within the GM and associated metabolites which contribute to CRS, ICANS and HLH and survival which are amenable to therapeutic targeting. For patients with follicular lymphoma, the investigators will assess if the GM affects the risk of disease progression and the need for systemic immuno-chemotherapy.

The ongoing collection of stool and blood samples from people with blood cancer or diagnosed with HLH will occur in a single centre, Nottingham University Hospitals NHS Trust. Samples will be used to study the effects of the host GM on toxicity, progression and survival. Stool and serum samples are planned to undergo shotgun metagenomics (microbiome profiling) and untargeted metabolomics. Multi-omics integration analysis will be conducted, including taxonomy, functional and metabolite analysis. Any remaining samples will, given patient permission, be kept for future ethically approved related studies, including potential downstream investigations such as organ-on-chip (gut, liver, brain), stool and serum mRNA analysis (RNA-seq) to identify downregulated targets, stool and blood non-coding RNA analyses, proteomics, epigenomics and glycomics as well as in vivo zebrafish and/or other animal studies. Stool and peripheral blood mononuclear cells can be co-cultured in primary cell lines or organ-on-chips (EMULATE) to mimic disease and to evaluate therapies. These studies may be carried out at the University of Nottingham, or be transferred to other researchers within and outside of the UK and other commercial institutions.

The project will continue, until 1st January 2040, but renewal for the study may occur after this. Any plans to cease the study will be notified to the REC at least two months prior with information detailing how we plan to dispose of any remaining samples and/or details of transfer to another area/site. The ongoing collection of blood and stool for translational studies is extremely valuable in facilitating research into the outcomes of immunotherapy for blood cancer and HLH.

Participant duration:

The patients actively participate in the study for a maximum of 56 days to allow serial sample collection.

Patients receiving immunotherapy (BiSp or CART) for blood cancer will have samples collected on at baseline (within two weeks up to day 0), day 3 (+/- 24 hours) and day 28 (+/- 24 hours) of treatment.

Patients diagnosed with HLH will have samples collected within 48 hours of diagnosis, and between days 7-10 and days 28-30 post diagnosis.

Patients diagnosed with follicular lymphoma will have samples collected within 30 days of diagnosis only. The end of the study will be the last blood and serum sample taken from the last participant. Laboratory analyses will continue for up to a further five years.

Recruitment Participants will be recruited from haematology clinics and wards within Nottingham University Hospitals NHS Trust. As HLH is a clinical emergency all patents are already admitted, and potential patients may be enrolled onto the study on the same day as diagnosis. Patients with blood cancer will be approached and consented during successive clinic appointments. The initial approach will be from a member of the patient's usual care team (which may include the investigator).

The investigator or their nominee, e.g. from the research team or a member of the participant's usual care team, will inform the participant or their nominated representative (other individual or other body with appropriate jurisdiction), of all aspects pertaining to participation in the study.

If needed, the usual hospital interpreter and translator services will be available to assist with discussion of the trial, the participant information sheets, and consent forms, but the consent forms and information sheets will not be available printed in other languages.

It will be explained to the potential participant that that entry into the trial is entirely voluntary and that their treatment and care will not be affected by their decision. It will also be explained that they can withdraw at any time but attempts will be made to avoid this occurrence. In the event of their withdrawal it will be explained that their data collected so far cannot be erased and we will seek consent to use the data in the final analyses where appropriate. Remaining tissue samples can be destroyed if the participant so wishes.

Standard of care patient diagnostics will be recorded by the haematology clinical and or research team for later correlation with findings, and will include:

1. Age, sex, ethnicity, body mass index medical history, Charlson co-morbidity score, concomitant medications including antibiotic/probiotics use and duration, and food frequency questionnaire.
2. Haematology, biochemistry and microbiology results, and biopsy/bone marrow biopsy reports.
3. Details of lymphoma including histology, prior therapies and any CAR-T cell product administered.
4. Adverse events (CRS/ICANs and grade) and use of antibiotics, tocilizumab and steroids.
5. Progression free and overall survival.

All participants will provide written informed consent. Should there be any subsequent amendment to the final protocol, which might affect a participant's participation in the trial, continuing consent will be obtained using an amended Consent form which will be signed by the participant.

Study procedures The participants are attending the hospital for treatment of their haematological disease as part of their routine clinical care. By taking part in this study participants are also asked to give up to three stool samples over time, and an extra three blood samples (up to 50mls) which will be added to already planned venesection. Blood samples will be taken by NHS staff in the clinic and wards.

Sample size and justification We estimate that approximately 100 patients per year will be eligible (BiSp ~25/year, CAR-T ~50/year, HLH ~4/year, indolent lymphoma 20/year) and up to 50 patients per year will be enrolled. As the study is hypothesis generating, there is no formal sample size calculation.

Bioinformatics analysis and integration of gut microbiota and metabolomics data sets, will be performed within the University of Nottingham, as well as being performed by potential collaborators and PhD students.

Sample Labelling Each participant will be assigned a trial identity code number for use on the samples, consent forms and other study documents and the electronic database. The documents and database will also use their initials (of first and last names separated by a hyphen or a middle name initial when available) and date of birth (dd/mm/yy).

Source documents Source documents shall be filed at the investigator's site and may include but are not limited to, consent forms, current medical records, laboratory results and records. A CRF may also completely serve as its own source data. Only trial staff as listed on the Delegation Log shall have access to trial documentation other than the regulatory requirements listed below.

Direct access to source data / documents Study documents, including progress notes and copies of laboratory and medical test results shall made be available at all times for review by the Chief Investigator, Sponsor's designee and inspection by relevant regulatory authorities.

Data Protection All staff and investigators involved with the study will endeavour to protect participants' rights to privacy and informed consent, and will adhere to the Data Protection Act, 2018. Only the minimum required information for the purposes of the study shall be collected. Documents will be held securely, in a locked room, or locked cupboard or cabinet. Access to the information will be limited to the study staff and investigators and relevant regulatory authorities (see above). Computer held data including the study database will be held securely and password protected. All data will be stored on a secure dedicated web server. Access will be restricted by user identifiers and passwords (encrypted using a one way encryption method).

Information about the study in the participant's medical records / hospital notes will be treated confidentially in the same way as all other confidential medical information.

Study conduct Study conduct may be subject to systems audit of the study files for inclusion of essential documents; permissions to conduct the study; CVs of study staff and training received; local document control procedures; consent procedures and recruitment logs; adherence to procedures defined in the protocol (e.g. inclusion / exclusion criteria, timeliness of visits); and equipment calibration logs. The Chief Investigator, or nominated designee, shall carry out a site systems audit at least yearly and an audit report shall be made to the study Sponsor.

Study data Monitoring of study data shall include confirmation of informed consent; source data verification; data storage and data transfer procedures; local quality control checks and procedures, back-up and disaster recovery of any local databases and validation of data manipulation. The Chief Investigator, or where required, a nominated designee, shall carry out monitoring of study data as an ongoing activity.

Record retention and archiving In compliance with the DH Research Governance Framework guidelines, the Human Tissue Act and in accordance with the University of Nottingham Code of Research Conduct and Research Ethics, the Chief Investigator will maintain all records and documents of the study. These will be retained for at least 7 years or for longer if required. If the responsible investigator is no longer able to maintain the study records, a second person will be nominated to take over this responsibility.

The study documents held by the Chief Investigator on behalf of the Sponsor shall be finally archived at secure archive facilities at the University of Nottingham. This archive shall include all study databases and associated meta-data encryption codes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 16-100 years
* A blood cancer or clinically confirmed HLH by H-score criteria

Exclusion Criteria:

* Known positive HIV, hepatitis B and/or hepatitis C serology (as laboratory not accredited to handle high-risk samples).
* Active communicable disease eg SARS-CoV-2, monkeypox.

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from haematology clinics and wards within Nottingham University Hospitals NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2039-12-31 (Estimated); Study Completion 2044-12 (Estimated)

PRIMARY OUTCOMES:
To collect blood and stool samples from patients with blood cancer and/or HLH to enable the study of the influence of the host immune system and gut microbiota on toxicity and survival. | The patients actively participate in the study for a maximum of 56 days to allow serial sample collection.
  The study aims to assess characteristic baseline signatures and/or dynamic changes within the immune system and gut microbiome/metabolome predicting toxicity, progression and survival adult patients with blood cancer or HLH. The study is exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Bishton, MBChB, MRCP, FRCPath, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Microbiome sequencing data will be made open access and uploaded to NCBI and related repositories.